CLINICAL TRIAL: NCT00183625
Title: The Effectiveness of Supplementing Supported Employment With Behavioral Skills Training
Brief Title: Supported Employment and Skills Training in Conjunction With Pharmacotherapy in Schizophrenia Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01MH041573 (NIH); R01MH041573 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2005-11

CONDITIONS: Schizophrenia
Keywords: Antipsychotic Agents; Employment
MeSH Terms: conditions — Schizophrenia | interventions — Palliative Care; Employment, Supported; Olanzapine; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Risperidone Plus Supported Employment (Active Comparator)
  Interventions: Behavioral: Individual Placement and Support (Supported Employment); Drug: Risperidone
- Olanzapine Plus Supported Employment (Active Comparator)
  Interventions: Behavioral: Individual Placement and Support (Supported Employment); Drug: Olanzapine
- Risperidone+Supported Employment+Skills (Active Comparator)
  Interventions: Behavioral: Individual Placement and Support (Supported Employment); Behavioral: Social Skills Training; Drug: Risperidone
- Olanzapine+Supported Employment+Skills (Active Comparator)
  Interventions: Behavioral: Individual Placement and Support (Supported Employment); Behavioral: Social Skills Training; Drug: Olanzapine

INTERVENTIONS:
Behavioral: Individual Placement and Support (Supported Employment)
Behavioral: Social Skills Training
  Arms: Olanzapine+Supported Employment+Skills; Risperidone+Supported Employment+Skills
Drug: Olanzapine
  Arms: Olanzapine Plus Supported Employment; Olanzapine+Supported Employment+Skills
Drug: Risperidone
  Arms: Risperidone Plus Supported Employment; Risperidone+Supported Employment+Skills

SUMMARY:
This study will compare employment support with behavioral skills training to employment support alone in schizophrenia patients taking either risperidone or olanzapine to determine which is more effective in helping the patients maintain a job.

DETAILED DESCRIPTION:
Schizophrenia is a severe mental disorder characterized by disorganized thoughts, difficulty concentrating, and hallucinations. Individuals with schizophrenia often experience reduced emotional, social, and occupational functioning. Data indicate that antipsychotic drug treatment and occupational training and support may be effective in helping people with schizophrenia maintain a stable job. Risperidone and olanzapine are antipsychotic drugs; participants in this study will be taking either risperidone or olanzapine for the duration of the study. This study will provide schizophrenia patients with employment support alone or with behavioral skills training to determine which combination is more effective in helping patients obtain and maintain a job.

At study entry, participants will undergo a clinical and diagnostic evaluation to determine the severity of their schizophrenia. Participants will be tapered off their regular medication for schizophrenia over 4 weeks. At the end of Week 4, they will be randomly assigned to receive either risperidone or olanzapine. Participants will then be assigned an Individual Placement and Support (IPS) specialist to assist them in finding a job. After participants secure a job, they will be randomly assigned to receive IPS either alone or with the Workplace Fundamentals Skills Training Module for 2 years. Participants' risperidone or olanzapine treatment will continue during this 2-year period. Participants will have clinic visits at study entry and Months 7, 12, and 24. At each visit, participants will complete questionnaires and will be interviewed about their schizophrenia symptoms and occupational functioning.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia
* Candidate for maintenance schizophrenia treatment
* Willing to initiate and continue risperidone or olanzapine therapy for the duration of the study

Exclusion Criteria:

* Any serious medical problems other than schizophrenia that would interfere with the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2000-06; Primary Completion 2005-06 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R. Marder, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - West Los Angeles Veterans Healthcare Center, Los Angeles, California
  - Greater Manchester Mental Health Center, Manchester, New Hampshire

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited at the Manchester Mental Health Center, Greater Los Angeles VA, and UCLA Semel Institute
Groups:
- Risperidone Plus Supported Employment; Risperidone + Supported Employment + Skills; Olanzapine + Supported Employment + Skills: Participants were randomized at baseline to risperidone or olanzapine and Individual Placement and Support with or without workplace fundamentals. The WIPS was not implemented until participant obtained a job.
- Olanzapine Plus Supported Employment: Individual Placement and Support plus Olanzapine. Participants were randomized at baseline to risperidone or olanzapine and Individual Placement and Support with or without workplace fundamentals. The WIPS was not implemented until participant obtained a job.
Period: Overall Study
Arm/Group | Risperidone Plus Supported Employment | Olanzapine Plus Supported Employment | Risperidone + Supported Employment + Skills | Olanzapine + Supported Employment + Skills
Started | 27 | 28 | 28 | 24
Obtained employment | 21 | 18 | 14 | 14
Completed | 9 | 10 | 9 | 10
Not Completed | 18 | 18 | 19 | 14
Not completed — Withdrawal by Subject | 18 | 18 | 19 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Risperidone Treatment | Olanzapine Treatment | Total
Number analyzed (Participants) | 55 | 52 | 214
Age, Continuous [Mean (Standard Deviation); unit: years]
  number analyzed (Participants) | 55 | 52 | 107
  (all) | 41.8 (10.4) | 42.2 (9.4) | 42.0 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  number analyzed (Participants) | 55 | 52 | 107
  Female | 10 | 9 | 19
  Male | 45 | 43 | 88

OUTCOME MEASURES:

1. Primary Outcome: Total Weeks Worked
Time Frame: 24 months
Population: Data were analyzed for work condition (IPS with or without WIPS) and not for medication (risperidone or olanzapine)
Measure: Mean (Standard Deviation); unit: Weeks
Groups:
- Individual Placement and Support (IPS): IPS alone for risperidone and olanzapine subjects
- Individual Placement and Support With Workplace Fundamentals: Olanzapine and Risperidone Patients included.
Arm/Group | Individual Placement and Support (IPS) | Individual Placement and Support With Workplace Fundamentals
Number analyzed (Participants) | 39 | 28
Weeks | 51.53 (31.15) | 41.37 (37.46)
Statistical Analysis 1: Comparison: Individual Placement and Support (IPS) vs Individual Placement and Support With Workplace Fundamentals; Test type: Superiority or Other; p = 0.66, Regression, Linear

2. Secondary Outcome: Body Mass Index
Description: Intent was to compare medication and not work group conditions. This was initially assessed at baseline and includes total time on either risperidone or olanzapine up to 18 months.
Time Frame: First 18 months of study
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | Risperidone Treatment | Olanzapine Treatment
Number analyzed (Participants) | 55 | 52
kg/m^2 | 29.21 (.99) | 30.4 (1.04)
Statistical Analysis 1: Comparison: Risperidone Treatment vs Olanzapine Treatment; Mixed effects regression of body mass index on medication group (risp or olanz), time (in days over first 18 months of study) and a group by time interaction with site and baseline timepoint indicators as covariates. The model included a random slope and intercept for time; Test type: Superiority or Other; p = .0176, Mixed Models Analysis — The p-value listed is for the medication by time interaction

ADVERSE EVENTS:
Arm/Group | Risperidone Treatment | Olanzapine Treatment
Serious Adverse Events (participants affected / at risk) | 16/55 | 12/52
Other Adverse Events (participants affected / at risk) | 0/55 | 0/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risperidone Treatment (N=55) | Olanzapine Treatment (N=52)
Hospitalization (Psychiatric disorders) | 16 (34) | 12 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No